CLINICAL TRIAL: NCT05589077
Title: Effectiveness of an Educational Intervention Tool Related to Nutritional Concerns in Physically Active Female Young Adults
Brief Title: Knowledge of Nutritional Concerns in Physically Active Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-1348
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-10

CONDITIONS: Nutritional Deficiency
Keywords: Female Athlete; Sport Nutrition; Patient Education
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: All participants will complete the same survey and engage in the same intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knowledge Assessment and Educational Intervention (Experimental): All participants will be asked to complete the pre-intervention survey assessing knowledge and confidence of female athlete nutritional concerns. Then participants will engage in an educational intervention on these same topics. Following the intervention, participants will repeat the same survey.
  Interventions: Behavioral: Education on Female Athlete Nutritional Concerns

INTERVENTIONS:
Behavioral: Education on Female Athlete Nutritional Concerns — Visual and audio information presented within the Qualtrics system will cover topics on the Female Athlete Triad, Relative Energy Deficiency in Sport, and eating disorders.

SUMMARY:
Purpose: The purpose of this study is to determine whether implementation of an educational tool for nutritional concerns in 18-25-year-old females who participate in sport increases their understanding of various nutritional concerns. By studying an educational tool geared towards nutritional concerns of the female athlete, clinicians can use the information to improve clinical practice and patient outcomes.

Procedure: Participants will be asked to complete a previously validated survey assessing knowledge of nutritional concerns of female athletes: the Female Athlete Triad, Relative Energy Deficiency in Sport, and eating disorders. The survey will be completed immediately pre- and post-receipt of the educational intervention. The intervention includes education on the previously mentioned nutritional concerns.

DETAILED DESCRIPTION:
The current study is a quasi-experimental study consisting of one virtual session on Qualtrics. Eligible participants (as determined via a screening questionnaire) will use a link to access the questionnaire online. The questionnaire will collect information on participant's demographic background. Then, participants compete a 37-item survey on nutritional concerns and rate their confidence in each answer. Participants were given a score of 1 if the answer was correct, and a score of -1 if the answer was incorrect. Corresponding to each Knowledge question was a Likert scale for confidence (i.e. "How confident are you in this response?"). Response options on the Confidence options ranged from 0 to 5, with 0 indicating "No confidence" and 5 indicating "Completely sure". The range of total scores for Knowledge ranged from -37 to +37 with +37 indicating greatest amount of knowledge. The total Confidence score was the sum of all confidence responses from each of the scored knowledge questions. The total number of Confidence points ranged from 0-148. A higher confidence score indicated greater confidence from the participant in their knowledge answers. Impact scores were also calculated to measure the total composite score of Knowledge plus Confidence to identify an increased understanding of all scores.

Impact scores will be calculated using the same procedure as Lodge et al. (2020): "The total points of impact score from the questionnaire range between +37 and -37. A percentage of impact can be calculated using the limits -37 to +37 of the impact score (range of 74 points). A score of 0 will have a percentage of 50%, a score of -37 will have a percentage of 0%, and a score of +37 will have a percentage of 100%. Each question has a score range between +1 and -1. One point is given for the correct answer and high confidence and one point is subtracted for the incorrect answer and high confidence. The score of the questions is reduced when the respondent has lower confidence in their answer. The scale of confidence corresponds to the following points for impact scoring: Confidence 4 = 1 point, Confidence 3 = 0.75 points, Confidence 2 = 0.5 points, Confidence 1 = 0.25 points, Confidence 0 = 0 points. For example, if the answer is correct with the lowest confidence (1), it is scored as 0.25. If the answer is incorrect with the lowest confidence (1), it is scored as -0.25. If the answer selected if "I don't know", or a confidence of zero (0) is selected, it is scored as zero. For questions of "choose all that apply" nature, each possible sub-answer is considered individually".1

Then, participants will engage in a 10-minute educational intervention. The intervention will cover all the information regarding nutritional concerns that were tested in the survey. Participants will repeat the same survey to test their knowledge and confidence in nutritional concerns. Lastly, participants will answer 10 follow-up questions.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-25
* Participate in organized sport

Exclusion Criteria:

* Must meet all inclusion criteria (no previous or current health concerns will exclude a participant from the study)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge Score | ~10 min for pre-test followed by ~10 min intervention followed by ~10 min post-test.
  Participants will be asked 37 questions in the survey assessing their knowledge on nutritional concerns. Each correctly answered question is worth 1 point and each incorrectly answered question is worth -1 point. The highest possible score a participant can receive is 37. The lowest possible score a participant can receive is -37. Higher scores indicate higher levels of knowledge.
Change in Confidence Score | ~10 min for pre-test followed by ~10 min intervention followed by ~10 min post-test.
  Corresponding to each Knowledge question was a Likert scale for confidence (i.e. "How confident are you in this response?"). Response options on the Confidence options ranged from 0 to 5, with 0 indicating "No confidence" and 5 indicating "Completely sure". The total Confidence score is the sum of all confidence responses from each of the scored knowledge questions. The total number of Confidence points ranged from 0-148. A higher confidence score indicates greater confidence from the participant in their knowledge answers. Higher scores indicate higher levels of confidence.
Change in Impact Score | ~10 min for pre-test followed by ~10 min intervention followed by ~10 min post-test.
  The score quantifies the correctness of an answer combined with the level of confidence. Each question has a score range between -1 and 1. The correctness of the answer and level of confidence in the answer produces the Impact score. One point is given for the correct answer and high confidence and one point is subtracted for the incorrect answer and high confidence. The score of the questions is reduced when the respondent has lower confidence in their answer. The scale of confidence corresponds to the following points for impact scoring: Confidence 4 = 1 point, Confidence 3 = 0.75 points, Confidence 2 = 0.5 points, Confidence 1 = 0.25 points, Confidence 0 = 0 points. The total Impact score is the sum of each question's score. Higher scores indicate both high levels of knowledge and confidence simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Woelffer, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Data will be made available from the PI upon request.

REFERENCES:
- [Background] Lodge MT, Ackerman KE, Garay J. Knowledge of Triad and RED-S in Female Cross-Country Athletes and Support Staff. J Athl Train. 2021 Jul 30. doi: 10.4085/1062-6050-0175.21. Online ahead of print. PMID 34329432